CLINICAL TRIAL: NCT02304562
Title: Umbilical Cord Blood-derived Mesenchymal Stem Cells in Regeneration of Sweat Glands and Body Repair
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xiaobing Fu, Academician, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHIN-PLAGH-ST-004
Record Dates: First submitted 2014-11-21; First posted 2014-12-02 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Sweat Gland Diseases
MeSH Terms: conditions — Sweat Gland Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- UCB Mesenchymal Stem Cells (Experimental): UCB Mesenchymal Stem Cells treatment of patients with skin injury
  Interventions: Biological: UCB Mesenchymal Stem Cells treatment

INTERVENTIONS:
Biological: UCB Mesenchymal Stem Cells treatment — reduce skin injury

SUMMARY:
Patients with skin injury treated with Umbilical Cord Blood-derived Mesenchymal Stem Cells,such as deep burn damaged sweat glands,Effectiveness of Umbilical Cord Blood-derived Mesenchymal Stem Cells in Regeneration of Sweat Glands and Body Repair is determined.

ELIGIBILITY:
Inclusion Criteria:

* Burn area:10-20％TBSA

Exclusion Criteria:

* Have influence on the speed of wound healing of patients with chronic diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events | 6 months
  Frequency and severity of Adverse Events

SECONDARY OUTCOMES:
Active and inactive lesion count | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: xiaobing FU, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Fu X, Qu Z, Sheng Z. Potentiality of mesenchymal stem cells in regeneration of sweat glands. J Surg Res. 2006 Dec;136(2):204-8. doi: 10.1016/j.jss.2005.03.024. Epub 2006 Oct 20. PMID 17056067